CLINICAL TRIAL: NCT01013324
Title: A Phase 2 Study of XL147 (SAR245408) in Subjects With Advanced or Recurrent Endometrial Carcinoma
Brief Title: Study of XL147 (SAR245408) in Advanced or Recurrent Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD11436; XL147-201 (Other: (Other study code))
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms
Keywords: endometrial cancer; endometrial carcinoma; carcinoma of the endometrium; cancer of the endometrium
MeSH Terms: conditions — Endometrial Neoplasms | interventions — XL147

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): All subjects will receive single-agent XL147 dosed daily
  Interventions: Drug: XL147 (SAR245408)

INTERVENTIONS:
Drug: XL147 (SAR245408) — dosed as capsules taken orally daily

SUMMARY:
There has not been any systemic therapy approved in the United States or in Europe for treating advanced or recurrent endometrial cancer (EC). This study will evaluate the safety and preliminary efficacy of XL147 in advanced or recurrent EC.

Constitutively active phosphatidylinositol-3 kinase (PI3K)/phosphatase and tensin homolog on chromosome 10 (PTEN) pathway signaling is common in EC and involved in the development and/or progression of the disease. PTEN deficiency and/or activating mutations/amplification in the PIK3CA gene that encodes the p110α catalytic subunit of PI3K have been frequently detected in EC patients. XL147 is a potent and highly selective inhibitor of the Class I PI3K family of lipid kinases. In addition, in vivo preclinical data have demonstrated that XL147 targets both proximal and distal signaling in the PI3K/PTEN pathway. Therefore, XL147 may have utility in the treatment of subjects with advanced or recurrent EC.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed diagnosis of EC (endometrioid, serous, clear cell adenocarcinoma, adenosquamous carcinoma, or mixed histology, any grade) that is advanced (ie, persistent, locally advanced) or recurrent, and is incurable by standard therapies and has received one platinum based chemotherapy regimen for EC.
* The subject is at least 18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The subject has at least one measurable lesion
* Tissue samples from archival or fresh tissue, or a tissue block of the subject's tumor
* The subject has adequate organ and marrow function
* The subject is capable of understanding the informed consent and complying with the protocol and has signed the informed consent document before any study-specific screening procedures or evaluations are performed.
* Sexually active subjects of childbearing potential and their partners must agree to use medically accepted methods of contraception during the course of the study and for 3 months after discontinuation of study drug.
* Subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* The subject has previously been treated with a selective PI3K inhibitor, mTOR inhibitor, or AKT inhibitor.
* The subject has uterine sarcomas (leiomyosarcoma), mixed Mullerian tumors, squamous carcinoma of the uterus, and/or adenosarcomas of the uterus.
* Certain restrictions on prior treatments apply
* The subject has not recovered from toxicity due to prior therapy to Grade ≤ 1 or to pre-therapy baseline (excluding alopecia and peripheral neuropathy).
* The subject has a known primary brain tumor or brain metastasis.
* The subject has any other diagnosis of malignancy or evidence of malignancy (except non-melanoma skin cancer or in situ carcinoma of the cervix) within 2 years before screening for this study.
* The subject has a diagnosis of uncontrolled diabetes mellitus or has a fasting plasma glucose > 160 mg/dL.
* The subject is currently receiving anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤ 1 mg/day is permitted).
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test results at screening that are above 1.3 x the laboratory upper limit of normal.
* The subject has uncontrolled, significant intercurrent illness
* The subject has a baseline corrected QT interval ≥ 470 ms.
* The subject is known to be positive for the human immunodeficiency virus (HIV). (Note: Baseline HIV screening is not required.)
* The subject is pregnant or breastfeeding.
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy as defined by overall response rate and progression-free survival (PFS) at 6 months | every 8-10 weeks
Safety of XL147 in the EC population | scheduled evaluations every 2-4 weeks

SECONDARY OUTCOMES:
Duration of response and PFS | every 8-10 weeks
Characterize pharmacokinetic and pharmacodynamic profiles of XL147 | at periodic visits not less than every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (10):
  - Investigational Site Number 1526, Newport Beach, California
  - Investigational Site Number 1532, Orlando, Florida
  - Investigational Site Number 1239, Augusta, Georgia
  - Investigational Site Number 1133, Boston, Massachusetts
  - Investigational Site Number 1325, Columbus, Ohio
  - Investigational Site Number 1434, Oklahoma City, Oklahoma
  - Investigational Site Number 1132, Abington, Pennsylvania
  - Investigational Site Number 1134, Philadelphia, Pennsylvania
  - Investigational Site Number 1142, Providence, Rhode Island
  - Investigational Site Number 1527, Dallas, Texas
- Belgium (3):
  - Investigational Site Number 3212, Kortrijk
  - Investigational Site Number 3211, Leuven
  - Investigational Site Number 3218, Wilrijk